CLINICAL TRIAL: NCT01117818
Title: A Randomized, Controlled, Parallel Group, Double-blind, Multi-center, Phase II Study to Assess the Clinical- and Immunological Activity,as Well as the Safety and Tolerability of Different Doses/Formulations of AFFITOPE AD02 Administered Repeatedly to Patients With Early Alzheimer's Disease
Brief Title: Clinical- and Immunological Activity, Safety and Tolerability of Different Doses / Formulations of AFFITOPE AD02 in Early Alzheimer's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Affiris AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AFF006; 2009-016504-22 (EudraCT Number)
Record Dates: First submitted 2010-04-19; First posted 2010-05-06 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- A: AFFITOPE AD02 (Active Comparator)
  Interventions: Biological: active: AFFITOPE AD02
- B: AFFITOPE AD02 (Active Comparator)
  Interventions: Biological: active: AFFITOPE AD02
- C: AFFITOPE AD02 (Active Comparator)
  Interventions: Biological: active: AFFITOPE AD02
- D: Placebo control (Active Comparator)
  Interventions: Biological: control: Placebo

INTERVENTIONS:
Biological: active: AFFITOPE AD02 — vaccination
  Other Names: AFFITOPE AD02
  Arms: A: AFFITOPE AD02; B: AFFITOPE AD02; C: AFFITOPE AD02
Biological: control: Placebo — vaccination
  Other Names: placebo; control
  Arms: D: Placebo control

SUMMARY:
This is a multiple vaccination study to find out if it is a safe treatment and what effects it has on the symptoms of early Alzheimer's disease in male and female patients aged 50 to 80 years. Approximately 40 study sites in Europe will be involved. Patients will be randomized to receive either AFFITOPE AD02 or placebo. Each patient's participation will last 1 year.

DETAILED DESCRIPTION:
AFFITOPE AD02 is a second generation AD immunotherapeutics targeting Aβ. Its active component is a synthetic peptide functionally mimicking the unmodified N-terminus of Aβ.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent capability
* Early AD, based on episodic memory deficit and hippocampal atrophy
* Age from 50 to 80, inclusive
* MMSE of 20+
* Brain magnetic resonance imaging scan consistent with the diagnosis of AD
* Stable doses of medications (cholinesterase inhibitors and memantine allowed)
* Caregiver able to attend all visits with patient

Exclusion Criteria:

* Significant neurological disease other than AD
* Major psychiatric illness
* Significant systemic illness
* Autoimmune disease
* Prior treatment with experimental immunotherapeutics for AD including IVIG
* Women of childbearing potential without birth control
* Contraindication for MRI scan

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 335 (Actual)
Dates: Start 2010-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
cognitive(ADAS-cog modified) and functional(ADCS-ADL modified) | 18 months

SECONDARY OUTCOMES:
cognitive(computerised test battery), global(CDR-sb), behavioral(NPI), biomarker (volumetric MRI) | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Dubois, Prof, Principal Investigator — Centre des Maladies Cognitives et Comportementales, Federation des maladies du systeme nerveux, Hoptial de la Salpetriere, Pavillon Paul Castaignes (Sous-sol), 47-83 Bd de l'Hopital, 75651 Paris Cedex 13
Locations (31):
- Austria (7):
  - Landeskrankenhaus Hall Gedächtnisambulanz, Hall in Tirol
  - LNK Wagner-Jauregg, Dept. of geriatrics, Linz
  - Christian Doppler Klinik, Univ. Klinik f. Neurologie, Salzburg
  - Studienzentrum der PROSENEX, Ambulatoriumbetriebsges.m.b.H an der Confraternität - Privatklinik Josefstadt, Vienna
  - MUW Klin. Pharmakologie und Klinik für Neurologie, Vienna
  - MUW, Klin.Abt.f. Biolog. Psychiatrie, Vienna
  - SMZ-Ost, Psychiatric Dep., Vienna
- Croatia (5):
  - Klinčki Bolnički Centar Rijeka, Klinika za Psihijatriju, Rijeka
  - Opća bolnica Varaždin, Klinika za Neurologiju, Varaždin
  - "BONIFARM" Poliklinika za kliničku farmakologiju i toksikologiju, Zagreb
  - Klinčki Bolnički Centar Zagreb (REBRO), Klinika za Neurologiju, Zagreb
  - Psihijatrijska Bolnica Vrapče, Zagreb
- Czechia (2):
  - University Thomayer Hospital, Prague
  - University Hospital Motol, Clinic of Neurology, Prague
- France (7):
  - CMRR Hôpital Pellegrin, Bâtiment USN Tastet Girard, Bordeaux
  - Hôpital Neurologique Pierre Wertheimer, Bron
  - Centre Hospitalier Universitaire (CHU) de Dijon, Dijon
  - Centre Mémoire de Ressources et de Recherche, Service de Neurologie, Montpellier
  - Hôpital de la Pitié-Salpêtrière, Paris
  - CHU de rennes Site Hôtel Dieu, Rennes
  - Hopital La Grave, Toulouse
- Germany (8):
  - Charite Universitätsmedizin Berlin, Klinik u. Hochschulambulanz f. Psychiatrie u. Psychotherapie, Berlin
  - Universitätsklinikum Hamburg-Eppendorf, Klinik für Psychiatrie und Psychotherapie, Hamburg
  - Arzneimittelforschung Leipzig GmbH, Studienzentrum, Leipzig
  - Zentralinstitut für Seelische Gesundheit, Abt. Gerontopsychiatrie, Mannheim
  - Klinik u. Poliklinik f. Psychiatrie u. Psychotherapie der TU München, Munich
  - Studienzentrum PD Dr. Steinwachs, Nuremberg
  - Klinikum Nürnberg Nord, Klinik f. Psychiatrie u. Psychotherapie, Nuremberg
  - NeuroPoint GmbH, Ulm/Donau
- Slovakia (2):
  - EPAMED, s.r.o., Košice
  - Psychiatric Hospital Michalovce, Michalovce